CLINICAL TRIAL: NCT01816256
Title: Screening for Asymptomatic Portal Vein Thrombosis and Portal Hypertension in Patients With Philadelphia Negative Myeloproliferative Neoplasms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MPN 12-01
Record Dates: First submitted 2013-01-14; First posted 2013-03-22 (Estimated); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Myeloproliferative Neoplasms (MPN); Polycythemia Vera (PV); Essential Thrombocythemia (ET); Myelofibrosis (MF)
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Screening tests (Other): This is a one arm study. All patients will receive two screening tests (Doppler ultrasound, upper gastrointestinal endoscopy).
  Interventions: Procedure: Upper gastrointestinal endoscopy and Doppler ultrasound

INTERVENTIONS:
Procedure: Upper gastrointestinal endoscopy and Doppler ultrasound — This is a one arm study. All patients will receive two screening tests (Doppler ultrasound, upper gastrointestinal endoscopy).

SUMMARY:
This study involves screening for portal vein thrombosis and portal hypertension in patients with Philadelphia negative myeloproliferative neoplasms (MPNs). These include polycythemia vera (PV), essential thrombocythemia (ET), and myelofibrosis.

Portal vein thrombosis and portal hypertension are serious complications that are often seen in myeloproliferative patients. These complications are usually diagnosed when patients become symptomatic, and are often already at an advanced stage. They can further progress to cause non-reversible damage to the liver, also called cirrhosis of the liver. As a result of this, patients often accumulate fluid in the abdomen which is ascites; and can develop swelling of veins in the lining of the esophagus known as varices. If untreated, varices have the risk of rupturing resulting in life-threatening bleeding. When diagnosed at an advanced stage, the treatment is usually supportive therapy and there are no treatments available at present which can reverse these conditions.

This study is looking at screening for these two conditions using Doppler ultrasound and upper gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* One of the three classical Philadelphia negative myeloproliferative neoplasms (polycythemia vera (PV), essential thrombocythemia (ET) and myelofibrosis (MF)) diagnosed according to WHO or International working group-Myelofibrosis research and treatment (IWG-MRT) criteria
* Palpable spleen length greater than 5 cm below the costal margin in MF (including primary MF or post-polycythemia vera MF (PPV-MF) post-polycythemia vera ET (PPV-ET)) or palpable spleen of any size in patients with PV or ET.
* Ability to understand and willing to sign a written consent form.
* Age 18 years or older at time of consent.

Exclusion criteria:

* Known history of portal vein thrombosis
* Known history of Budd-chairi syndrome
* Known history of oesophageal varices
* Known history of cirrhosis from any cause
* Known history of active bleeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-05; Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Incidence of asymptomatic portal vein thrombosis (PVT) and/or portal hypertension (PHTN) in patients with Philadelphia negative myeloproliferative neoplasms (MPNs) | 6 years

SECONDARY OUTCOMES:
Identify the patient, disease and treatment related risk factors associated with PVT and PHTN | 6 years
Comparison of survival and number of patients with leukemic transformation in patients with or without asymptomatic PVT/PHTN | 8 years

OTHER OUTCOMES:
Identify any genetic markers or biomarkers associated with asymptomatic PVT and PHTN | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gupta, MD, FRCP, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario